CLINICAL TRIAL: NCT02560636
Title: Phase I Study of Hypofractionated Radiotherapy and Anti-PD1 Antibody (Pembrolizumab) in the Treatment of Advanced Bladder Cancer
Brief Title: Pembrolizumab in Muscle Invasive/Metastatic Bladder Cancer
Acronym: PLUMMB
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Institute of Cancer Research, United Kingdom (Other); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CCR 4255
Record Dates: First submitted 2015-09-21; First posted 2015-09-25 (Estimated); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Invasive Bladder Cancer
Keywords: Muscle Invasive; Metastatic; Advanced
MeSH Terms: conditions — Neoplasm Metastasis | interventions — pembrolizumab; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Dose level 1a (Experimental): Radiotherapy: 24Gy in 6f Pembrolizumab: 100mg
  Interventions: Drug: Pembrolizumab; Radiation: Radiotherapy
- Dose level 1b (Experimental): Radiotherapy: 24Gy in 6f Pembrolizumab: 200mg
  Interventions: Drug: Pembrolizumab; Radiation: Radiotherapy
- Dose level 2a (Experimental): Radiotherapy: 24Gy in 4f Pembrolizumab: 100mg
  Interventions: Drug: Pembrolizumab; Radiation: Radiotherapy
- Dose level 2b (Experimental): Radiotherapy: 24Gy in 4f Pembrolizumab: 200mg
  Interventions: Drug: Pembrolizumab; Radiation: Radiotherapy
- Dose level 3a (Experimental): Radiotherapy: 30Gy in 5f Pembrolizumab: 200mg
  Interventions: Drug: Pembrolizumab; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab - Trial Treatment
  Other Names: MK-3475/pembrolizumab (KEYTRUDA®)
Radiation: Radiotherapy — Radiotherapy

SUMMARY:
PLUMMB is an phase I trial to investigate the safety, tolerability and effectiveness of an immunotherapy drug called Pembrolizumab used in combination with radiotherapy. The study will also investigate two different doses of pembrolizumab, starting at 100mg (through an intravenous drip) and increasing to 200mg for the next cohort of patients, if the first dose is well tolerated. The patients suitable for this study will be: Group A those with locally advanced bladder cancer or Group B patients whose cancer has spread from the bladder (metastatic bladder cancer).

Treatment in the PLUMMB trial will start with a pembrolizumab 2 weeks prior to starting a course of 4 - 6 weeks radiotherapy. Treatment with pembrolizumab will then be given every three weeks. Patients in Group A will then continue to take pembrolizumab for up to a year unless they have disease progression or unacceptable side effects in the meantime. Patients in Group B will continue taking pembrolizumab for as long as needed until they have disease progression or unacceptable side effects.

Patients will be seen every 3 weeks during treatment and every 3-6 months thereafter. CT scans will be done every 3 months during treatment and as per usual care (usually 6 monthly) after the treatment has finished. Patients in Group A will also have a cystoscopy (camera test) to look into the bladder 3 months after they finish radiotherapy. This is standard care and would be the same for patients not on a research study.

DETAILED DESCRIPTION:
1. Risk and burden for patients

   Patients in this study have cancer that often proves hard to control with standard care. The early phase nature of this study means that the intervention may not have any benefit for patients who take part in the study. However, they will still receive the standard treatment of radiotherapy. Throughout the study, any patients who have significant side effects from the trial drug will be withdrawn from the trial and will still be eligible to receive standard care. The study itself carries a number of potential burdens:
   * Experimental nature of the study drug. The drug stimulates the immune system to produce more proteins that will attack the tumour cells. It is thought that this will be selective for tumour cells; however it is possible that effects on normal tissues may cause side effects. These risks will be managed as much as possible by regular (3 weekly) clinical assessments as a hospital outpatient, by experienced clinicians while having the study treatment. Comprehensive assessments for safety will be carried out including more intensive monitoring with blood tests.
   * Burden of frequent hospital visits and tests. Participants in this study must attend hospital frequently for safety reasons to check for any toxicity of the study treatment. Blood tests (more than usual), clinical examination and urine tests are part of the safety assessment.
   * Additional investigations may be carried out as part of the study, for research purposes for which consent will be sought form the patient, such as additional blood samples and additional scans (CT thorax, abdomen and pelvis).
2. Phase 1 trial of Pembrolizumab: Patients will be carefully monitored for toxicity throughout the trial. A phase I trial has already been conducted to determine the maximum tolerated dose (MTD) of pembrolizumab in bladder cancer. To date no MTD has been defined and the maximum dose tested showed acceptable toxicity and positive effects on reducing tumour size. This study will assess two dose levels of pembrolizumab: 100mg and 200mg and differing radiotherapy doses (24-30Gy in 4-6f). Dose escalation will only occur if the current cohort have shown no signs of unacceptable toxicity at 6 weeks after completing radiotherapy.
3. Recruitment

   Participants will be offered information about this study by their clinical teams if they are considered to meet the entry criteria and express interest in taking part in an experimental study. It will be made clear that the study is experimental in nature and that there will not necessarily be a therapeutic benefit from taking part in the study. It will also be made clear that, should patients decide not to take part their future care will not be affected. Patients will be given sufficient time and information to make an informed decision about entering the trial, and not less than 24 hours; all patients entering the trial will give written informed consent. Inclusion and exclusion criteria for this study are standard for a phase 1 trial of a new oncology drug.
4. Confidentiality

   Patients will be linked to a unique identifier the code for which will be held on a password protected database held only by the study team. Blood samples, tumour sample processing and other data analysis will take place at the laboratories of Royal Marsden and Institute of Cancer Research in London or Sutton. Sample processing will take place using the study number only. No other patient identifiable information will be available on study samples. Investigators will have access to patient identifiable information on password protected NHS hospital notes and databases only.
5. Conflict of Interest

   Patients may be recruited to the study by those involved in their prior clinical care. The investigators do not expect conflict of interest between research and healthcare duties for a number of reasons: patients must give their full informed consent before entering the study, specifically regarding the unknown efficacy of the study drug and the intensive nature of the study. Those patients who do not continue in the study will maintain a relationship with the clinical team if required for symptom control. At the end of the study, patients will be able to access the results if they wish, through the Royal Marsden Website or contact the study team directly.
6. Use of tissue samples in future research

If participants give their consent, any leftover blood or tissue samples which are not required for this study will be stored for future unspecified research in line with the human tissue act regulations. Access and use of samples for research purposes will require appropriate ethical approval. Future researchers will not be able to identify individual patients from their biobank data, demographic and clinical information will be available.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed invasive bladder.carcinoma (T2-4,N0-3,M0-1).
2. Be willing and able to provide written informed consent for the trial.
3. Be ≥ 18 years of age on day of signing informed consent.
4. Have measurable disease based on RECIST 1.1. , or, in group A, disease assessable by cystoscopic assessment.
5. Have consented to analysis of tissue from an archival tissue sample
6. Have a performance status of 0-1 on the ECOG Performance Scale.
7. Planned for hypofractionated radiotherapy
8. Demonstrate adequate organ function as defined in table 2 (please see protocol) all screening blood tests should be performed within 10 days of confirmation of eligibility.
9. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to confirmation of study eligibility. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
10. Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
11. Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy if their partner has childbearing potential (as defined by not being surgically sterilized or have not been free from menses for > 1 year).

Exclusion Criteria:

The subject must be excluded from participating in the trial if the subject:

1. Is currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of treatment.
2. Previous pelvic radiotherapy, history of inflammatory bowel disease or other conditions that would in the opinion of the investigator would preclude the safe administration of pelvic radiotherapy.
3. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy (>dose equivalent to 10mg of Prednisolone/day) or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
4. Has had a prior monoclonal antibody within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
5. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent or therapy.

   * Note: Subjects with ≤ Grade 2 neuropathy or chemotherapy induced alopecia/nail changes are an exception to this criterion and may qualify for the study.
   * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
6. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, localized prostate cancer (≤T2 ≤ Gl3+4) or in situ cervical cancer that has undergone potentially curative therapy. Patients may have received treatment for previous urothelial malignancy.
7. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment.
8. Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Subjects with vitiligo or resolved childhood asthma/atopy would be an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Subjects with hypothyroidism stable on hormone replacement or Sjorgen's syndrome will not be excluded from the study.
9. Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
10. Has an active infection requiring systemic therapy.
11. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
12. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
13. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
14. Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
15. Has a known history of Human Immunodeficiency Virus (HIV).
16. Has known clinical history of Hepatitis B or Hepatitis C .
17. Has received a live vaccine within 30 days prior to the first dose of trial treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2016-06-06 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2028-07-30 (Estimated)

PRIMARY OUTCOMES:
Establishing the maximum tolerated dose (MTD) | up to 36 months
  Establishing the maximum tolerated dose (MTD) that can be safely combined with hypofractionated radiotherapy to the bladder in the absence of dose limiting toxicity (DLT) by assessing adverse events in the patient population.
Measurement of the rates of toxicity | 6 weeks after the last fraction of radiotherapy has been administered
  Adverse events will be graded and assessed by CTCAEv4.

SECONDARY OUTCOMES:
Measurement of the percentage of patients experiencing late grade 2+ and 3+ toxicity | 6 weeks and one day following the completion of radiotherapy until the 28 days after the patients last dose of Pembrolizumab
  Late grade 2+ and 3+ adverse events will be assessed by CTCAEv4.
Measuring rates of tumour response to treatment. | 3 months after completion of radiotherapy
  Determining the proportion of patients treated with the combination of Pembrolizumab and radiotherapy with local control of their bladder cancer (based on cystoscopy and/or diffusion weighted MRI) via RECIST.
Measurement of progression free and overall survival rate | Long term survival followup (reported at 2 years)
  Measurement of progression free and overall survival rate

OTHER OUTCOMES:
Measurement of progression-free survival in patients with no PD-1/PDL-1 expression vs high levels of PD-1/PDL-1 in their tumour | 36 months
  Measurement of progression-free survival in patients with no PD-1/PDL-1 expression vs high levels of PD-1/PDL-1 in their tumour
Report the proportion of patients free of grade 2 or higher toxicity | 3 and 6 months postradiotherapy completion
  Adverse events will be graded and assessed by CTCAEv4.
Report the proportion of patients with complete or partial response in non-irradiated metastases | 3 and 6 months
  Report the proportion of patients with complete or partial response in non-irradiated metastases measured via RECIST.

CONTACTS AND LOCATIONS:
Overall Officials: Professor Robert Huddart, Study Director — Royal Marsden NHS Foundation Trust
Locations (1):
- NIHR Biomedical Research Centre at RM and ICR (https://www.cancerbrc.org/), Sutton, United Kingdom

REFERENCES:
- [Derived] Tree AC, Jones K, Hafeez S, Sharabiani MTA, Harrington KJ, Lalondrelle S, Ahmed M, Huddart RA. Dose-limiting Urinary Toxicity With Pembrolizumab Combined With Weekly Hypofractionated Radiation Therapy in Bladder Cancer. Int J Radiat Oncol Biol Phys. 2018 Aug 1;101(5):1168-1171. doi: 10.1016/j.ijrobp.2018.04.070. Epub 2018 May 4. PMID 30012528